CLINICAL TRIAL: NCT04620161
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Proof of Concept Study to Assess the Efficacy, Safety and Tolerability of Pradigastat in Patients With Functional Constipation
Brief Title: A Proof of Concept Study of Pradigastat in Patients With Functional Constipation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anji Pharma (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANJ908C2101
Record Dates: First submitted 2020-10-21; First posted 2020-11-06 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Functional Constipation
Keywords: Pradigastat; Proof of Concept; Functional Constipation
MeSH Terms: interventions — pradigastat

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind and placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pradigastat Tablets 20mg (Experimental): The patients in this arm will receive one tablet a day of Pradigastat 20mg and one tablet a day of Pradigastat 40mg matching placebo
  Interventions: Drug: Pradigastat Tablets 20mg; Drug: Pradigastat Tablets 40mg matching Placebo
- Pradigastat Tablets 40mg (Experimental): The patients in this arm will receive one tablet a day of Pradigastat 40mg and one tablet a day of Pradigastat 20mg matching placebo
  Interventions: Drug: Pradigastat Tablets 40mg; Drug: Pradigastat Tablets 20mg matching Placebo
- Placebo (Placebo Comparator): The patients in this arm will receive one tablet a day of Pradigastat 20mg matching placebo and one tablet a day of Pradigastat 40mg matching placebo
  Interventions: Drug: Pradigastat Tablets 20mg matching Placebo; Drug: Pradigastat Tablets 40mg matching Placebo

INTERVENTIONS:
Drug: Pradigastat Tablets 20mg — 20mg, once daily, oral administration
  Other Names: ANJ908 20mg
  Arms: Pradigastat Tablets 20mg
Drug: Pradigastat Tablets 40mg — 40mg, once daily, oral administration
  Other Names: ANJ908 40mg
  Arms: Pradigastat Tablets 40mg
Drug: Pradigastat Tablets 20mg matching Placebo — once daily, oral administration
  Other Names: ANJ908 20mg matching Placebo
  Arms: Placebo; Pradigastat Tablets 40mg
Drug: Pradigastat Tablets 40mg matching Placebo — once daily, oral administration
  Other Names: ANJ908 40mg matching Placebo
  Arms: Placebo; Pradigastat Tablets 20mg

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of pradigastat 20 and 40 mg as compared to placebo in patients with Functional Constipation.

DETAILED DESCRIPTION:
This multicenter, randomized, placebo-controlled, double-blind study is designed to demonstrate the efficacy, safety and tolerability of pradigastat relative to placebo across 2 doses (20 and 40 mg) for up to 6 weeks (4-week treatment, 2-week Follow-up) in patients with Functional Constipation.

The primary endpoint is the change from baseline in the number of weekly spontaneous bowel movement (SBM), the key secondary endpoint is the change from baseline in the number of weekly complete spontaneous bowel movement (CSBM).An SBM is defined as a stool not induced by rescue medication, whereas a CSBM is defined as an SBM associated with a sensation of complete evacuation.

Summary of Protocol Amendments:

* Original Protocol: 06 January 2020
* Amendment 1: 30 July 2020 (Reason: To respond Health Authority requests)
* Amendment 2: 05 March 2021 (Reason: Sponsor decided to amend the protocol. Key changes: inclusion/exclusion criteria, criteria for Discountinuation from study/Discontinuation from Study Medication, adding the instruction for evaluating and managing diarrhea AEs. )

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Male and female patients aged 18 to 70 years of age, inclusive.
3. Patients with FC as defined by the ROME IV diagnostic criteria for FC.

   Diagnostic criteria for FC*:
   * Must include 2 or more of the following:

     1. Straining during more than one-fourth (25%) of defecations
     2. Lumpy or hard stools (Bristol Stool Form Scale 1 or 2) more than one-fourth (25%) of defecations
     3. Sensation of incomplete evacuation more than one-fourth (25%) of defecations
     4. Sensation of anorectal obstruction/blockage more than one-fourth (25%) of defecations
     5. Manual maneuvers to facilitate more than one-fourth (25%) of defecations (such as digital evacuation, or support of the pelvic floor)
     6. Fewer than 3 SBMs per week
   * Loose stools are rarely present without the use of laxatives
   * Insufficient criteria for irritable bowel syndrome (IBS). *Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis.
4. Patient has less than 3 SBMs/week within 2 weeks prior to the Screening Visit.
5. Patient has completed a colonoscopy with no clinically significant findings which meet other exclusion criteria within 12 months prior to Screening or at the Screening Visit.
6. Patient must agree that after the Visit 2 (Run-in Visit) they will discontinue any prohibited medications, laxatives (prescription and over-the-counter), supplemental fibers, or traditional medicine taken for abdominal symptoms or constipation as defined per protocol except the rescue medication, provided by the study site and following the Investigator's instructions for its use. Patient should not take rescue medication (bisacodyl) on the calendar day before and the calendar day of the start of the Treatment Period (Visit 3). If the wash-out criteria are not achieved on Visit 3, the Visit could be postponed once.
7. Patient must agree to use and comply with the diet guidance provided in applicable Chronic Constipation Treatment Guideline starting after the Screening Visit and during the study until End of Study.
8. Ability of patient to swallow tablets.
9. A co-operative attitude and ability to perform all study related procedures and to correctly use the diary.

Exclusion Criteria:

1. Patient with history of surgical resection of stomach, gallbladder, small intestine, large intestine, and bariatric surgery (excluding resection of appendicitis and benign polyp).
2. Patient with history or current affection of inflammatory bowel disease (Crohn's disease or ulcerative colitis) and celiac disease.
3. Patient with diagnosis of IBS (constipation, diarrhea, or mixed).
4. Patient with history or current ischemic colitis.
5. Patient currently with infectious enteritis or enterocolitis. Patients with asymptomatic diverticulosis, diagnosed during the colonoscopy can be enrolled, unless previous history of diverticulitis.
6. Patient currently with hyperthyroidism or hypothyroidism (unless adequately treated), or patients who have a thyroid-stimulating hormone outside of the laboratory reference range at Visit1.
7. Patient with apparent mechanical obstruction (ie, patient with ileus caused by hernia).
8. Patient has a structural abnormality of the GI tract or a disease or history of a condition that can affect GI motility.
9. Patient has ever had any of the following diseases or conditions that can be associated with constipation: pseudo-obstruction, colonic inertia, megacolon, megarectum, bowel obstruction, descending perineum syndrome, solitary rectal ulcer syndrome, and systemic sclerosis.
10. Patient currently affected by constipation due to anorectal disease, affecting the anorectal area such as anal fissure, anorectal fistulas, hemorrhoidal disease Grade III and IV, and bleeding hemorrhoids.
11. Patient currently has both unexplained and clinically significant alarm symptoms (lower GI bleeding, rectal bleeding or heme-positive stool, iron-deficiency anemia or any unexplained anemia, or weight loss) or systemic signs of infection or colitis.
12. Patient currently affected by drug-induced constipation.
13. Patient with constipation due to other organic disease.
14. Patient currently affected by active peptic ulcer (ie, disease that is not adequately treated or stable with therapy).
15. In the case of a female, the one currently affected by endometriosis or uterine adenomyosis.
16. Patient with uncontrolled severe depression, anxiety, or any eating disorder considered by the Investigator to influence drug evaluation.
17. Patient has a potential central nervous system cause of constipation (eg, Parkinson's disease, spinal cord injury, and multiple sclerosis.).
18. Patients with uncontrolled and unstable diabetes mellitus with reported episodes of hypoglycemia within 1 year prior to Screening or history of diabetic neuropathy.
19. Patient with history of abuse of drug or alcohol within 1 year before consent acquisition, or with current abuse.
20. Patient with history of or current diagnosis of any cancer (except for nonmelanoma skin cancer which has been removed) diagnosed less than 5 years prior to Screening. Patients with cancer in full remission more than 5 years after diagnosis are acceptable.
21. Patient with major surgery or any other condition that may require use of narcotic drugs or general anesthesia within 60 days of Screening and during the study.
22. Any clinically significant abnormality identified by physical examination, electrocardiogram (ECG) or laboratory tests, which in the judgment of the Investigator would compromise the patient's safety or successful participation in the clinical study, or any of the following laboratory findings:

    1. Male hemoglobin < 12 g/dL (< 120 g/L) and female hemoglobin < 10 g/dL (< 100 g/L) at Screening.
    2. Male serum creatinine ≥ 1.5 mg/dL and female serum creatinine ≥ 1.4 mg/dL, or creatinine clearance ≤ 60 mL/min based on calculation using the Cockcroft-Gault formula: ([140-age in years] × weight in kg)/(72 × [creatinine in mg/dL]). For women, multiply result by 0.85.
    3. Active liver disease and/or significant abnormal liver function defined as aspartate aminotransferase > 2 × upper limit of the normal (ULN) and/or alanine aminotransferase > 2 × ULN and/or total bilirubin > 1.5 × ULN.
    4. Patient with stool blood positive at Screening.
23. Patient currently affected by clinically significant cardiovascular disease, respiratory disease, kidney disease, hepatic disease, GI disease (excluding FC), hematology disease, endocrine disease, hemorrhagic disease, or neural/mental disease or other disease or condition that might, in the judgment of the Investigator, place the patients at undue risk or potentially compromise the results of interpretation of the study results.
24. Patient with history of drug allergy to any active or inactive ingredient of pradigastat.
25. Patients who are vegetarian or vegan.
26. Pregnant or nursing (lactating) women.
27. Women of childbearing potential, unless they are using effective methods of contraception during study.
28. Male, who are attempting to naturally father a child or donate sperm.
29. Patients who have received an investigational drug within 30 days or 5 half-lives (whichever is greater) prior to the Screening Visit.
30. Patients participating to another clinical study at any time during this study. Studies that require consent only to store data and that do not require Follow-up are not considered to be observational or interventional and are exempted from this exclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of pradigastat in changing the weekly spontaneous bowel movement (SBM) number compared with placebo in patients with functional constipation (FC) | Week 4
  Number change from baseline in the weekly SBM at Week 4

SECONDARY OUTCOMES:
Efficacy of pradigastat in changing the weekly complete spontaneous bowel movement (CSBM) number compared with placebo in patients with FC | Week 4
  Number change from baseline in the weekly CSBM at Week 4
Safety assessed by incidence of Adverse Events | Each visit through Week 4
  Safety assessed by incidence of Adverse Events
Efficacy of pradigastat in changing the responder rate compared with placebo in patients with FC | From baseline to every week until Week 4
  Weekly response rate for SBM
Change in weekly score for overall assessment of constipation symptoms and accompanied GI symptoms | From baseline to every week until Week 4
  Change in weekly score for overall assessment of constipation symptoms and accompanied GI symptoms (Weekly score includes 10 questions with the range of the total score from 10 to 68, and lower scores mean a better outcome.)
Trough pradigastat plasma concentrations | Week 1 and Week 4
  Mean plasma pradigastat concentration

CONTACTS AND LOCATIONS:
Overall Officials: Dan Meyers, M.D., Study Chair — Anji Pharma
Locations (25):
- United States (5):
  - Advanced Clinical Research-Meridian, Meridian, Idaho
  - Evanston Premier Healthcare Research, Evanston, Illinois
  - Jubilee Clinical Research, Las Vegas, Nevada
  - Long Island Gastrointestinal Research Group LLP, New York, New York
  - PMG Research of Charleston, Mt. Pleasant, South Carolina
- China (20):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Quanzhou First Hospital, Quanzhou, Fujian
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangsu University, Suzhou, Jiangsu
  - Yangzhou First People's Hospital, Yangzhou, Jiangsu
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Siping Central People's Hospital, Siping, Jilin
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hopsital, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital Affiliated to Medical College of Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang